CLINICAL TRIAL: NCT03326180
Title: Study of Peri-Articular Anaesthetic for Replacement of the Knee
Acronym: SPAARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Hemant Pandit, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OR16/88494; 2016-003154-32 (EudraCT Number); 197936 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2017-10-11; First posted 2017-10-31 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine (EXPAREL) (Experimental): 266mg/20ml EXPAREL mixed with 80ml 0.9% normal saline and 100mg/20ml 0.5% plain bupivacaine hydrochloride. Administered as a single dose intra-operatively by periarticular infiltration.
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine hydrochloride
- Bupivacaine hydrochloride alone (Active Comparator): 100ml 0.9% normal saline mixed with 100mg/20ml 0.5% plain bupivacaine hydrochloride.
  Administered as a single dose intra-operatively by periarticular infiltration.
  Interventions: Drug: Bupivacaine hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — 266mg/20ml vial of EXPAREL
  Other Names: EXPAREL
  Arms: Liposomal bupivacaine (EXPAREL)
Drug: Bupivacaine hydrochloride — 100mg/20ml 0.5% bupivacaine hydrochloride. Branded or generic, must be plain (cannot contain adrenaline/epinephrine)
  Other Names: Marcain

SUMMARY:
The clinical and cost effectiveness of peri-articular liposomal bupivacaine plus bupivacaine hydrochloride compared with bupivacaine hydrochloride alone for post-operative recovery after knee replacement surgery: A multi-centre, patient-blinded, randomised controlled trial.

DETAILED DESCRIPTION:
The trial design is a patient-blinded multi-centre, active comparator, randomised controlled two-arm parallel group superiority trial of liposomal bupivacaine plus bupivacaine hydrochloride versus bupivacaine alone for post-operative pain in patients undergoing knee replacement surgery.

Patients will be randomised in a 1:1 ratio. The randomised controlled trial (RCT) design is robust and reduces any potential bias. Patients will be blinded as to which treatment they receive. Blinding of patients is possible as they will be under general anaesthetic for their knee replacement surgery at the time of the drug administration. Blinding of surgeons, who administer the medication and outcome assessors was not necessary as the primary outcome is a patient reported outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary knee replacement, including both total knee replacement (TKR) or unicompartmental knee replacement (UKR), for end stage osteoarthritis
* American Society of Anaesthesiologists (ASA) Grade I to III
* Participant is willing and able consent for themselves
* Male or Female, aged 18 years or above
* In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

* Allergy or intolerance to amide type local anaesthetics
* Objective evidence of nerve damage in the affected lower limb.
* Rheumatoid arthritis
* Any other significant disease, disorder or condition which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the results of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 6 months.
* Participants who have significant cognitive impairment or language issues
* Contra-lateral knee replacement within the trial or within 12 months prior to randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 (QoR-40) | Change in score between 0, 24, 48 and 72 hours post-operatively
  A 40-item instrument which encompass most aspects of a good quality of recovery after surgery. Consists of five clinically relevant dimensions:
  1. Physical comfort (12 items)
  2. Emotional state (9 items)
  3. Physical independence (5 items)
  4. Psychological support (7 items)
  5. Pain (7 items).
  The QoR-40 has a possible score of 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Cumulative 0-10 pain Visual Analogue Score (VAS) | Cumulative score at 0, 24, 48 and 72 hours post-operatively
  Cumulative daily pain score at rest.
  A 10 point scale where 0 = no pain, 5 = moderate pain and 10 = worst possible pain.

SECONDARY OUTCOMES:
Mean 0-10 pain Visual Analogue Score (VAS) | 0, 24, 48 and 72 hours post-operatively
  Mean daily pain score at rest.
  A 10 point scale where 0 = no pain, 5 = moderate pain and 10 = worst possible pain.
Opioid consumption | Change in consumption between 0, 24, 48 and 72 hours post-operatively
  Cumulative consumption
Fitness for discharge (as per routine clinical care) | Assessed at 0, 24, 48 and 72 hours post-operatively
  Against pre-defined criteria. Patients would be considered fit for discharge when they meet the following criteria: Ability to mobilize independently; pain score less than or equal to 3mm on a 10 VAS; ability to straight leg raise and ability to bend knee to 90 degrees
Oxford Knee Score (OKS) | Change in score between baseline, 72 hours, 6 weeks, 6 months, 1 year post-operatively
  Functional outcome using validated, patient reported questionnaire
American Knee Society Score (AKSS) | Change in score between baseline, 72 hours, 6 weeks, 6 months, 1 year post-operatively
  Functional outcome using validated, patient reported questionnaire
EuroQol 5 Dimension scale | Change in score between baseline, 72 hours, 6 weeks, 6 months, 1 year post-operatively
  Validated patient reported quality of life questionnaire
Health economics | Change in cost utility between baseline, 6 weeks, 6 months, 1 year post-operatively
  Cost utility analysis
Serious Adverse Events (SAE) | Within 30 days of surgery
  Specifically cardiovascular or wound complications

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Pandit, Principal Investigator — University of Leeds
Locations (11):
- United Kingdom (11):
  - The Royal Orthopaedic Hospital, Birmingham
  - Chapel Allerton Hospital, Leeds
  - Pilgrim Hospital, United Lincolnshire Hospitals NHS Trust, Lincoln
  - The Whittington Hospital, London
  - Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry
  - Rotherham Hospital, Rotherham
  - King's Mill Hospital, Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Torbay Hospital, Torquay
  - Pinderfields Hospital - Mid Yorkshire, Wakefield
  - Yeovil District Hospital, Yeovil
  - York Teaching Hospital, York

IPD SHARING:
Plan to Share IPD: No